CLINICAL TRIAL: NCT07297290
Title: Effect of Metformin Use on Weight Loss in Obese, Non-diabetic People
Brief Title: Effect of Metformin Use on Weight Loss in Obese, Non-diabetic People (MOWRI)
Acronym: MOWRI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Of Nigeria Teaching Hospital (Network)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Ifeyinwa Nnakenyi, Consultant Chemical Pathologist and Metabolic Physician, University Of Nigeria Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024CWR-LMIC-981332295
Record Dates: First submitted 2025-09-01; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity and Cardiovascular Risk; Insulin Resistance; Obesity (Body Mass Index >30 kg/m2)
Keywords: Obesity; Metformin use; Weight loss; Non-diabetic
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded Pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Metformin 500mg extended release tablets taken once daily to a maximum dose of 1500mg daily
  Interventions: Drug: Metformin
- Control arm (Placebo Comparator): Identical-looking placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500mg extended release tablets taken to a maximum of 1500mg once daily
  Arms: Treatment arm
Drug: Placebo — Starch-based, identical looking placebo
  Arms: Control arm

SUMMARY:
Obesity is a chronic disease of global public health concern, contributing to cardiovascular disease, type 2 diabetes and certain cancers. Currently approved anti-obesity drugs and surgery are expensive and not readily available in Nigeria.

Metformin, approved for type 2 diabetes, has been shown to promote weight loss among obese patients in high income countries. However, metformin's effects have not yet been demonstrated in Black African populations, which may have different genetic and environmental predispositions to obesity and to the effect of metformin. This blinded, placebo-controlled, randomized trial is determining the effect of metformin on weight loss, cardiovascular disease risk and insulin resistance in Black Nigerians.

ELIGIBILITY:
Inclusion Criteria:

* • Obesity (defined as body mass index ≥ 30kg/m2),

  * Fasting plasma glucose (<7.0mmol/L)
  * No medical treatment for weight control in the previous 12 months
  * No participation in a current clinical trial

Exclusion Criteria:

* • Obesity (defined as body mass index ≥ 30kg/m2),

  * Fasting plasma glucose (<7.0mmol/L)
  * No medical treatment for weight control in the previous 12 months
  * No participation in a current clinical trial

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Metformin on body weight change | 24 months
  Determine percent change in body weight in kilograms and height in meters which will be combined to report BMI in kg/m2 among the treatment arm and compared to the control arm.
Effect of Metformin on Cardiovascular risk | 24 months
  Determine percent change in the 10 year Framingham risk score for cardiovascular disease among the treatment arm and compare with the control arm.
Effect of Metformin on insulin resistance in non-diabetics | 24 months
  Determine percent change in the insulin resistance indices using Homeostatic model assessment (HOMA) among the treatment arm and compare to the control arm.
Effect of metformin on waist circumference change | 24 months
  Determine the percent change in waist circumference measured in cm at baseline and final readings among the treatment arm and compared to the control arm.
Effect of metformin on waist-to-hip circumference change | 24 months
  Determine the percent change in waist circumference measured in cm, and hip circumference measured in cm, which will be combined to report waist-to-hip circumference ratio change among the treatment arm and compared to the control arm.

SECONDARY OUTCOMES:
Safety of Metformin extended release tablet taken daily | 24 months
  Determine the incidence of adverse effects at grade 3 or higher level using the Adverse Effect questionnaire when dosage of less than or equal to 1500mg of Metformin X extended release tablet is taken daily.
Percent drug compliance to Metformin extended release taken once daily. | 24 months
  Determine the percent drug compliance to administered Metformin extended release tablets, determined by count of actual number of drug tablets administered over count of what was expected to have been administered, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: IFEYINWA D NNAKENYI, MD, Principal Investigator — University Of Nigeria Teaching Hospital
Locations (2):
- Nigeria (2):
  - Pathology Facility, Enugu, Enugu State
  - University of Nigeria Teaching Hospital, Enugu, Enugu State

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form, Non-identifiable patient measurements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available after publishing of the research work likely from 1 Jan 2029 for 5 years (31 Dec 2033)
Access Criteria: The research institution, the research funders, potential collaborators and funders.